CLINICAL TRIAL: NCT06317805
Title: Randomized Trial Comparing Efficacy and Safety of Initial Triple Therapy Including Parenteral Treprostinil to Initial Double Oral Therapy in Pulmonary Arterial Hypertension (PAH) Group I Patients (TripleTRE)
Brief Title: Initial Triple Therapy Including Parenteral Treprostinil vs Initial Double Oral Therapy in PAH Group I Patients
Acronym: TripleTRE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Collaborators: ANOVA CRO s.r.o. (Unknown); PharmaLex Belgium (Unknown); Aixial s.r.o. (Unknown); GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREV1-10P.401; 2023-504351-26-01 (EU CTIS Number)
Record Dates: First submitted 2024-02-20; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: intermediate-high risk; intermediate-low risk with severe hemodynamic impairment
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-arm, open-label, low-interventional, phase IV, multi-centre clinical trial comparing efficacy and safety of initial triple therapy including parenteral treprostinil to initial double oral therapy (background therapy with endothelin receptor antagonist - ERA and phosphodiesterase type-5 inhibitor - PDE-5i) by proportion of patients achieving low risk status according to the simplified four-strata risk-assessment tool from week 24 up to 48 weeks in 110 (55/group) treatment-naïve adult intermediate-high risk or intermediate-low risk patients with severe hemodynamic impairment with pulmonary arterial hypertension (PAH) (group I).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial triple therapy (Experimental): Assigned treatment: double oral (background therapy consisting of 1 endothelin receptor antagonist ERA and 1 phosphodiesterase type-5 inhibitor PDE-5i) with subcutaneous (SC)/intravenous (IV) treprostinil on top
  Interventions: Drug: Generic treprostinil sodium + Standard of Care (Double Oral); Drug: Standard of Care - Double Oral
- • Initial double therapy (Active Comparator): double oral (background therapy consisting of 1 endothelin receptor antagonist ERA and 1 phosphodiesterase type-5 inhibitor PDE-5i)
  Interventions: Drug: Standard of Care - Double Oral

INTERVENTIONS:
Drug: Generic treprostinil sodium + Standard of Care (Double Oral) — Treprostinil (prostacyclin analogue) solution for continuous subcutaneous (SC) or intravenous (IV) infusion (1 mg/ml; 2.5 mg/ml; 5 mg/ml; 10 mg/ml in 10 mL glass vial) will be administered by an infusion pump system and up-titrated to ≥40 ng/kg/min or to the maximum tolerated dose within 24 weeks. Further up-titration shall be performed until trial completion according to the discretion of the investigator.
  Other Names: Trisuva, Tresuvi, Treposa, Treprostinil Orpha-Devel, Treprostinil Amomed, Treprostinil OrPha, Treposuvi
  Arms: Initial triple therapy
Drug: Standard of Care - Double Oral — All patients will receive standard of care double oral background treatment consisting of one Phosphodiesterase type 5 inhibitor (i.e., tadalafil or sildenafil) and one Endothelin Receptor Antagonist (i.e. ambrisentan, bosentan or macitentan)

SUMMARY:
TripleTRE investigates the effect of initial triple combination therapy (oral endothelin receptor antagonist (ERA) + oral phosphodiesterase tyüe-5 inhibitor (PDE-5i) + parenteral treprostinil) compared to double oral therapy (oral ERA + oral PDE-5i) in pulmonary arterial hypertension (PAH) patients (group I) with intermediate-high risk or patients with intermediate-low risk with severe hemodynamic impairment at baseline in a prospective, randomized, unblinded setting with scope of increasing evidence for optimization of therapy concepts in PAH.

The effect of initial triple combination therapy vs initial double oral therapy (standard of care (SoC)) will be measured by primary endpoint: (non)response to the assigned treatment.

DETAILED DESCRIPTION:
TripleTRE is prospective, randomized, two-arm, open-label, low-interventional, phase IV, multi-centre clinical trial comparing efficacy and safety of initial triple therapy including parenteral treprostinil to initial double oral therapy (standard of care (SoC)) by proportion of patients achieving low risk status according to the simplified four-strata risk-assessment tool from week 24 up to 48 weeks in 110 (55/group) treatment-naïve adult intermediate-high risk or intermediate-low risk participants with severe hemodynamic impairment with pulmonary arterial hypertension (PAH) (group I). Severe hemodynamic impairment is defined in current European Society of Cardiology (ESC)/European Respiratory Society (ERS) Guidelines as at least one of following conditions: mean right atrial pressure (RAP) ≥ 20 mmHg, cardiac index (CI) < 2.0 L/min, stroke volume index (SVI) < 31 mL/m2 and/or pulmonary vascular resistance (PVR) ≥ 12 WU. Risk status will be assessed with the simplified four-strata risk-assessment tool as per ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension (2022).

TripleTRE will be performed in adult participants with a confirmed diagnosis of idiopathic PAH (IPAH), hereditary PAH (HPAH), drug and toxin-induced PAH (DPAH), PAH associated with Connective Tissue Disease (PAH-CTD) and PAH with corrected congenital heart disease (PAH-CHD).

Participants will be randomized to one of the two treatment arms in 1:1 ratio. All patients will start with double oral background medication (endothelin receptor antagonist (ERA) and phosphodiesterase type-5 inhibitor (PDE-5i)). Choice of double oral drug combination underline the discretion of the investigator and applicable treatment guidelines. In both treatment arms all drugs (i.e., background medication in double oral group, background medication and parenteral treprostinil in initial triple group) will be initiated within 3 weeks after randomization. Patients randomized to treprostinil arm will receive training on infusion pump and medication after that investigational medicinal product will be handed out. All patients will be handed out diaries for documentation of treprostinil dose and used vials.

Primary objective of TripleTRE is to investigate the effect of initial triple combination therapy compared to initial double oral therapy on risk status. The effect of initial triple combination therapy vs initial double oral therapy (SoC) will be measured by primary endpoint: (non)response to the assigned treatment, whereas therapy responders/non-responders are defined as:

1. Therapy-responder: achievement of low-risk status between week 24 and week 48
2. Therapy-non-responder:

   1. pulmonary hypertension (PH) related deterioration to high-risk status, lung transplantation or death between week 12 and week 48 and/or
   2. additional medication or change of initial PH specific medication due to unsatisfactory efficacy between week 12 and week 48 and/or
   3. low risk status not achieved up to week 48

Risk status is assessed with the simplified four-strata risk-assessment tool as per ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension (2022).

Commonly used variables such as hemodynamics, echocardiogram (ECHO) and time to clinical worsening will be evaluated as secondary endpoints. In addition, the emPHasis-10 questionnaire will be used as disease specific and validated patient-reported outcome tool for PAH patients. The European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) will be used as general patient-reported outcome tool independent from disease.

TripleTRE trial is organized as a low-intervention trial consistent with definition in Clinical Trial Regulation (Regulation (EU) No 536/2014). Participants will not undergo any invasive examinations or laboratory evaluations, diagnostic or monitoring procedures specifically for the purposes of this trial that would expose them to increased risk compared to standard of care. Trial-related procedures as well as the frequency of assessments are in alignment with ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension (2022) and are not expected to pose additional risks to patients.

Planned trial duration per patient is minimum 12 weeks and maximum 48 weeks with up to 10 visits depending on achievement of therapy responder (i.e., low risk status) or therapy non-responder status. The visits 2 and 3 can be performed on phone. Other visits will be performed on-site. The trial will only be conducted in countries where ERA and PDE-5i treatments are standard of care and treprostinil is available to patients. At the end of trial, patients will be treated according to routine medical care at the PH expert centers receiving locally reimbursed medications. Approximately 10 countries and 20 sites are planed.

Statistical considerations:

The complete statistical analysis plan (SAP) was finalized before first patient in (FPI) in meaning of first act of recruitment. A one-sided Boschloo exact test at 2.5% significance level will be used to test the following primary hypothesis:

H0: Proportion of patients achieving low risk status (therapy responders) between week 24 and week 48 after baseline in the initial Triple treatment group is less or equal to the proportion of patients achieving low risk status between week 24 and week 48 after baseline in the initial Double oral treatment group.

The null hypothesis will be rejected if the 97.5% CI of the difference of proportions of therapy responders (triple minus double) is greater than 0.

To account for the variable time on treatment of therapy responders, a secondary sensitivity analysis will be performed by comparing the median time to the achievement of the low-risk status between the treatment groups.

Further sensitivity and subgroup analyses are defined in detail the statistical analysis plan (SAP) including the handling of missing values.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any trial-mandated procedure
* Male or female ≥ 18 and ≤ 70 years of age
* Symptomatic treatment-naïve PAH patients (group I) with confirmed diagnosis of one of the following subgroups:

  * idiopathic pulmonary arterial hypertension (IPAH)
  * hereditary pulmonary arterial hypertension (HPAH)
  * Drug and toxin-induced pulmonary arterial hypertension (DPAH)
  * PAH associated with Connective Tissue Disease
  * PAH with corrected congenital heart disease 4. Intermediate-high risk patients rated acc. the simplified four-strata risk-assessment tool or intermediate-low risk with severe hemodynamic impairment as defined in current PH guidelines i.e., mean right atrial pressure (RAP) ≥ 20 mmHg, cardiac index (CI) < 2.0 L/min, stroke volume index (SVI) < 31 mL/m2 and/or pulmonary vascular resistance (PVR) ≥ 12 WU
* Right Heart Catheterization (RHC) meeting all the following criteria:

  * Mean pulmonary arterial pressure (mPAP) > 20 mmHg
  * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg
  * PVR > 2 Wood Units
* Women of childbearing potential must not be pregnant or lactating, must perform regular pregnancy tests, if sexually active, agrees to continue to use reliable method(s) of contraception until study completion

Exclusion Criteria:

* PAH patients (group I) belonging to one of the following subgroups:

  * Schistosomiasis
  * HIV infection
  * Portal hypertension
  * Diffuse systemic sclerosis
  * Uncorrected congenital heart disease including uncorrected systemic-to-pulmonary shunts
* Any PAH-specific drug therapy in the past 3 months
* Patients responding to vasoreactivity testing with calcium channel blockers (CCB)
* Post-capillary PH and left heart disease
* Known or suspected pulmonary veno-occlusive disease (PVOD)
* Any PH due to lung disease
* Any disorder of the respiratory system expressed by Diffusing Capacity of Lung for Carbon Monoxide (DLCO) <40% and a noticeable imaging result (e.g., CT) and (Total Lung Capacity) TLC <60% and (Forced Expiratory Volume) FEV1 <70% by plethysmography (a pulmonary function test)
* Patients with need of ambulatory or long-term oxygen therapy
* Electrocardiogram (ECG) with Fridericia's corrected QT interval (QTcF) > 480 msec at screening
* Body mass index (BMI) > 35 (kg/m2)
* Age > 70 years
* History of restrictive, constrictive or congestive cardiomyopathy, atrial septostomy, any symptomatic coronary disease events within 6 months, severe uncontrolled arterial hypertension, acutely decompensated heart failure and myocardial infarction within 30 days, significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease, chronic systemic hypotension, unstable angina pectoris, permanent/persistent atrial fibrillation and/or need for pacemaker
* Patients with acute anemia with hemoglobin (Hb) values <11g/dL
* Cerebrovascular accident within 3 months
* Documented severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3× upper limit of the normal range (ULN) accompanied by aspartate aminotransferase (AST) > ULN and/or Child-Pugh Class C
* Documented renal insufficiency with Glomerular Filtration Rate (GFR) <30 ml/min
* Patients with untreated sleep apnea
* Patient with other cardiovascular, liver, renal, hematologic, gastrointestinal (including active gastrointestinal ulcer), immunologic, endocrine (e.g., uncontrolled diabetes), metabolic, or central nervous system disease and acute bleeding and injuries (e.g., intracranial hemorrhage) that, in the opinion of the investigator, may adversely affect the safety of the patient and /or efficacy of the therapy or significantly limit the lifespan (< 12 months)
* Patients with major surgery in the last 12 months
* Known history of alcohol abuse
* Treatment of a a cytochrome P450 (CYP)2C8 enzyme inducer (e.g., rifampicin) ≤ 28 days and/or treatment of a CYP2C8 enzyme inhibitor (e.g., gemfibrozil) ≤ 28 days
* Treatment with another investigational drug (planned, or taken ≤ 12 weeks)
* Hypersensitivity to any of the trial treatments or any excipient of their formulations
* Pregnancy, breastfeeding, or intention to become pregnant during the trial
* Any other significant disease or disorder which, in the opinion of the investigator, may put the patients at risk when participating in the trial
* Any factor or condition likely to affect protocol compliance of the patient, as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients achieving (non-)response status to the assigned treatment in terms of achievement of low-risk status | between week 12 and week 48 from baseline (BL)
  1. Therapy-responder: achievement of low-risk status between week 24 and week 48
  2. Therapy-non-responder:
     1. PH related deterioration to high-risk status, lung transplantation or death between week 12 and week 48 and/or
     2. additional medication or change of initial PH specific medication due to unsatisfactory efficacy between week 12 and week 48 and/or
     3. low risk status not achieved up to week 48 Risk status is assessed with the simplified four-strata risk-assessment tool as per PH guidelines.

SECONDARY OUTCOMES:
Change in hemodynamic parameters by means of right heart catheterization (RHC) - PVR | at week 24 from baseline (BL)
  Pulmonary Vascular Resistance (PVR) measured in WU
Change in hemodynamic parameters by means of right heart catheterization (RHC) - mPAP | at week 24 from baseline (BL)
  Mean pulmonary arterial pressure (mPAP) measured in mmHg
Change in hemodynamic parameters by means of right heart catheterization (RHC) - mRAP | at week 24 from baseline (BL)
  Mean right atrial pressure (mRAP) measured in mmHg
Change in hemodynamic parameters by means of right heart catheterization (RHC) - CI | at week 24 from baseline (BL)
  Cardiac index (CI) measured in liters per minute per square meter
Change in hemodynamic parameters by means of right heart catheterization (RHC) - CO | at week 24 from baseline (BL)
  Cardiac output (CO) measured in liters per minute
Change in hemodynamic parameters by means of right heart catheterization (RHC) - RAP | at week 24 from baseline (BL)
  Right atrial pressure (RAP) measured in mmHg
Change in right heart structure and function assessed by echocardiography - TAPSE/sPAP | at week 24 from baseline (BL)
  RV-PA coupling estimated by the ratio of tricuspid annular plane systolic excursion by pulmonary artery systolic pressure (TAPSE/sPAP)
Change in right heart structure and function assessed by echocardiography - RVEDA | at week 24 from baseline (BL)
  RV end-diastolic area (RVEDA) measured in square centimeters
Change in right heart structure and function assessed by echocardiography - RVESA | at week 24 from baseline (BL)
  RV end-systolic area (RVESA) measured in square centimeters
Change in right heart structure and function assessed by echocardiography - RVFAC | at week 24 from baseline (BL)
  RV fractional area change (RVFAC) calculated in %
Change in right heart structure and function assessed by echocardiography - RA | at week 24 from baseline (BL)
  Right Atrium (RA) area in square centimeters
Change in right heart structure and function assessed by echocardiography - Pericardial effusion | at week 24 from baseline (BL)
  Pericardial effusion assessment will be done and rated as yes/no
Time to achievement of low-risk status | time from baseline (BL) up to week 48
  Time from baseline to achievement of low-risk status assessed by the simplified four-strata risk-assessment tool
Rate of change of risk status | between baseline and week 48
  by means of the simplified four-strata risk-assessment tool categorizing patients in low (1), intermediate-low (2), intermediate-high (3) and high risk (4) based on the outcome in WHO FC class assessment, 6MWD and BNP/NT-proBNP
Change in the number of low-risk criteria based on the French PH Network Registry (FPHR) risk assessment tool | between baseline and week 24
Change in REVEAL 2.0 risk score | between baseline and week 24
  REVEAL Registry Risk Score 2.0 for Pulmonary Arterial Hypertension (PAH) predicts survival in patients with pulmonary arterial hypertension.
  It classifies patients in 3 risk groups:
  * Low: REVEAL score ≤6 meaning a predicted 1-year survival of ≥94%
  * Intermediate: REVEAL score 7-8 meaning a predicted 1-year survival of 70% to <94%
  * High: REVEAL score ≥9 meaning a predicted 1-year survival of <70%
Rate of change in WHO-FC | between baseline and week 48
Rate of change in 6MWD | between baseline and week 48
Rate of change in NT-proBNP/BNP levels | between baseline and week 48
Total number of clinical worsening(s) | between baseline and week 48
  where clinical worsening is defined as:
  * PAH related death (including all deaths where PAH cannot be excluded as cause) and lung transplantation due to PAH
  * PH-related hospitalization
  * Post baseline (screening visit) decrease in 6MWD by 15%
  * Post baseline (screening visit) worsening of WHO FC
Overall and transplant free survival | between baseline and week 48
Rate of change in quality of life - emPHasis-10 | between baseline and week 48
  Emphasis meaning something of special importance or significance. Please translate using the most appropriate term. The PH in emPHasis represents the condition Pulmonary Hypertension. The number 10 refers to the number of items in the questionnaire.
  This questionnaire is designed to determine how Pulmonary Hypertension (PH) affects patient's life. It refers to how PH affects or the impact that PH has on the patient's life.
Rate of change in quality of life - EQ-5D-5L | between baseline and week 48
  The EQ-5D-5L questionnaire consists of 2 parts - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. It should be noted that the numerals 1-5 have no arithmetic properties and should not be used as a cardinal score.

OTHER OUTCOMES:
Safety outcomes: | between baseline and week 48
  1. Number of Adverse events (AE) and Adverse reactions (ADR)
  2. Number of Serious Adverse events (SAE) and Serious Adverse Drug Reactions (SADR)
  3. Number of Suspected unexpected serious adverse reactions (SUSAR)

CONTACTS AND LOCATIONS:
Locations (19):
- Austria (2):
  - Ordensklinikum Linz, Linz
  - Medical University Vienna, Vienna
- Czechia (2):
  - Fakultní Nemocnice Olomouc, Olomouc
  - Všeobecná fakultní nemocnice v Praze, Prague
- France (2):
  - Hôpital Bicêtre-- Assistance Publique Hopitaux de Paris, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (3):
  - DRK Kliniken Berlin Westend, Berlin
  - University Hospital Carl Gustav Carus of Technical University Dresden, Dresden
  - Universitätsmedizin Greifswald, Greifswald
- Hungary (2):
  - Gottsegen National Cardiovascular lnstitute, Budapest
  - Medical University of Szeged, Szeged
- Sapienza University of Rome, Rome, Italy
- Poland (2):
  - John Paul II Hospital Krakow, Krakow
  - Fryderyk Chopin Hospital in European Health Centre Otwock, Otwock
- Centro Hospitalar Lisboa Norte - Santa Maria University Hospital, Lisbon, Portugal
- Romania (2):
  - Emergency Institute for Cardiovascular Diseases Prof. Dr. C.C.Iliescu, Bucharest
  - Emergency Clinical County Hospital of Targu Mures, Târgu Mureş
- Spain (2):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No